CLINICAL TRIAL: NCT00410267
Title: A Randomized Prospective Double - Masked Controlled Trial Comparing Ketorolac Tromethamine 0.4% and Prednisolone Acetate 1% in Reducing Post-Selective Laser Trabeculoplasty Anterior Chamber Flare and Cells
Brief Title: Trial Comparing Ketorolac Tromethamine 0.4% & Prednisolone Acetate 1% in Reducing Post-SLT Anterior Chamber Flare & Cells
Status: Terminated | Type: Observational
Why Stopped: low recruitment
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 0511006
Record Dates: First submitted 2006-12-11; First posted 2006-12-12 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2008-01

CONDITIONS: Postoperative Complications; Inflammation; Glaucoma, Open-Angle
Keywords: glaucoma; Post operative from selective laser trabeculoplasty
MeSH Terms: conditions — Postoperative Complications; Inflammation; Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
Selective laser trabeculoplasty (SLT) is a new alternative to anti-glaucoma medications for the treatment of primary open angle glaucoma. After SLT, many patients experience mild to moderate inflammation inside the eye - specifically in the front chamber of the eye (the part in front of the colored part of the eye). This mild front chamber reaction is typically treated with anti-inflammatory agents such as corticosteroids and nonsteroidal anti-inflammatory agents (NSAIDs). Some physicians do not use these agents as they feel they may interfere with the way the laser works to treat glaucoma. Topical (applied to the surface) corticosteroids can cause an increase in the pressure of the eye (intraocular pressure or IOP), cataract formation, or a possible increase in infection with long-term use. These side effects have not been reported to occur with NSAIDs, which are effective in controlling pain after SLT and reducing signs of inflammation such as irritation, swelling, tenderness, and soreness.

This research study will compare an NSAID, ketorolac tromethamine 0.4% (Acular LS), with a corticosteroid, prednisolone acetate 1% (Pred Forte), and with a placebo, which contains no active medicine (Refresh Tears). Ketorolac tromethamine 0.4%, prednisolone acetate 1%, and Refresh Tears are all FDA (Food and Drug Administration) approved for use in inflammation after surgery.

DETAILED DESCRIPTION:
Selective laser trabeculoplasty (SLT) is a new alternative to anti-glaucoma medications for the treatment of primary open angle glaucoma. After SLT, many patients experience mild to moderate inflammation inside the eye - specifically in the front chamber of the eye (the part in front of the colored part of the eye). This mild front chamber reaction is typically treated with anti-inflammatory agents such as corticosteroids and nonsteroidal anti-inflammatory agents (NSAIDs). Some physicians do not use these agents as they feel they may interfere with the way the laser works to treat glaucoma. Topical (applied to the surface) corticosteroids can cause an increase in the pressure of the eye (intraocular pressure or IOP), cataract formation, or a possible increase in infection with long-term use. These side effects have not been reported to occur with NSAIDs, which are effective in controlling pain after SLT and reducing signs of inflammation such as irritation, swelling, tenderness, and soreness.

This research study will compare an NSAID, ketorolac tromethamine 0.4% (Acular LS), with a corticosteroid, prednisolone acetate 1% (Pred Forte), and with a placebo, which contains no active medicine (Refresh Tears). Ketorolac tromethamine 0.4%, prednisolone acetate 1%, and Refresh Tears are all FDA (Food and Drug Administration) approved for use in inflammation after surgery.

To date, there is no study that proves that any one of the three study medications is better than the others for care after SLT. We plan to compare the effect of these anti-inflammatory drops in participants after selective laser trabeculoplasty to see if one works better at helping lower the pressure inside the eye after SLT or whether participants would do just as well with non-medicated eye drops. We will also see how well these drops reduce any potential discomfort and swelling that arise.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with open angle glaucoma at the University of Pittsburgh Medical Center (UPMC) Glaucoma Clinic.
* Able to provide written informed consent to participate.
* Must be between the ages of 18 - 95.
* Patients in which further IOP lowering by SLT is necessary in the opinion of the treating physician.

Exclusion Criteria:

* Patients with eye surgery in the prior six months.
* Patients with prior or current use of topical or systemic corticosteroids or NSAIDs.
* Patients with pre-existing anterior chamber inflammation.
* Patients with known sensitivity to any of the study medications.
* Due to the age range and the disease entity, special patient populations such as children or pregnant women will not be enrolled in this study.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2006-02; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Noecker, MD, Principal Investigator — University of Pittsburgh; Joel S Schuman, MD, Study Chair — University of Pittsburgh
Locations (1):
- University of Pittsburgh (UPMC Eye Center), Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No